CLINICAL TRIAL: NCT00545519
Title: A Phase I Study Of Thymoglobulin In Patients With Relapsed Or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-0946
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Relapsed Or Refractory Multiple Myeloma
Keywords: Multiple Myeloma; Thymoglobulin
MeSH Terms: conditions — Multiple Myeloma | interventions — thymoglobulin; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 1 (Experimental): Thymoglobulin 2.0 mg/kg over 8 hours on day 1 and over 6 hours on days 2-4.
  Interventions: Drug: thymoglobulin
- Dose Level 2 (Experimental): Thymoglobulin 3.0 mg/kg over 8 hours on day 1 and over 6 hours on days 2-4.
  Interventions: Drug: thymoglobulin
- Dose Level 3 (Experimental): Thymoglobulin 4.0 mg/kg over 8 hours on day 1 and over 6 hours on days 2-4.
  Interventions: Drug: thymoglobulin

INTERVENTIONS:
Drug: thymoglobulin
  Other Names: Vidaza

SUMMARY:
To determine the maximum tolerated dose and dose limiting toxicity of thymoglobulin in multiple myeloma patients.

To determine the overall response rate (CR+PR) of patients with relapsed or refractory multiple myeloma treated with Thymoglobulin.

To determine the time to response, duration of response, and time to progression and overall survival of patients treated with Thymoglobulin.

To determine the safety and tolerability of Thymoglobulin in these patients.

To assess the changes in lymphocyte apoptosis and apoptotic signaling in treated patients.

DETAILED DESCRIPTION:
Increasingly, upregulation of antiapoptotic proteins have been implicated in the pathogenesis and in the development of chemotherapy resistance in multiple myeloma. Therapeutic interventions that target the apoptotic pathway in myeloma are attractive targets to treat resistant disease. Dexamethasone triggers apoptosis via the release of Smac (second mitochondria-derived activator of caspase) leading to the activation of caspase-9 and caspase-3.37 The proteasome inhibitor bortezomib blocks signal transduction pathways mediated by NF-κB including the regulation of antiapoptotic genes such as TRAF1 and 2 (TNF receptor-associated factors) and cIAP (cellular inhibitor of apoptosis) and BCLXL.

Two independent investigators have established the activity of thymoglobulin in multiple myeloma cells from cell lines and patients.38,39 Thymoglobulin has been shown to induce apoptosis via distinct mechanisms in multiple myeloma cells.40 This action appears to be mediated by interactions with surface markers including CD80, CD38, CD40 and CD45. This appears to stimulate apoptosis via cathepsin and caspase pathways.39 By targeting different aspects of the apoptotic process, Thymoglobulin may provide a mechanism to overcome drug resistance in multiple myeloma.

Normal bone marrow B-cells, activated B cells and plasma cells have been shown to undergo apoptosis in a concentration dependent manner with rATG. The rATG has been shown to bind to B cells and this binding competitively inhibits several B cell specific monoclonal antibodies. The apoptosis can be inhibited by specific pathway inhibitors to caspases, cathepsin B and lysosomal cysteine proteases, indicating that each of these pathways is stimulated by thymoglobulin exposure. 18

Thymoglobulin at high concentrations binds complement resulting in direct cell lysis of lymphocytes.22 Anti-thymocyte globulins induce B cell apoptosis and do so preferentially to myelomonocytic and T-cell lines.41,42 Both myeloma cell lines and primary myeloma cells from patient bone marrow aspirates undergo apoptosis after exposure to thymoglobulin, as might be expected based on the apoptotic affect on B-cell lineages.38 Additionally both sets of cells undergo opsonization when complement is added in vitro. This demonstrates that thymoglobulin can induce myeloma cell kill by a number of methods and thus would be less susceptible to tumor resistance. The thymoglobulin binding sites have been assessed by competitive binding with monoclonal antibodies. Thymoglobulin binds competitively and specifically to IgG, HLA-ABC, HLA-DR, CD16, CD32, CD64, CD19, CD20, CD27, CD30, CD38, CD40, CD52, CD80, CD95, CD126, and CD138. Only IgG, CD16, CD64, and CD80 are not competitively bound. The apoptosis in primary cells can be inhibited by blocking the caspase, cathepsin D, or cathepsin B & D pathways. Zand et al also compared apoptotic response for five different lots of thymoglobulin. All lots apoptotic curves were overlapping over the range of 1-120 mcg/ml, demonstrating that very little lot to lot variation exists.43 This would be expected since each lot is derived from the combined sera of multiple immunized rabbits and thus individual differences in response for each rabbit would be mitigated. This may not be the case with lots of ATGAM each derived from a single horse. Each lot of thymoglobulin is already depleted of antibodies to red blood cells, has viruses inactivated and is tested for lymphocytotoxicity prior to release. The consistency demonstrated by Zand et al is consistent with the lack of observed variation in potency noticed in the greater than 20 years of clinical experience with this medication.

Together, these data provide a rational for the clinical use of Thymoglobulin in multiple myeloma. As a result, we propose a dose escalation, phase I, open-label study of Thymoglobulin in patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma diagnosed by standard criteria.
2. Measurable levels of monoclonal protein in serum (> 0.5 g/dL) or urine (> 0.2 g/24 hr).
3. At least 2 prior therapies for multiple myeloma with documented evidence of progression on the most recent treatment.
4. Age 18 years or older.
5. ECOG performance status <= 2.
6. Acceptable organ and marrow function as defined below:

   * Hemoglobin > 8 gm/dL
   * Absolute neutrophil count > 1,000/mm3
   * Platelets > 50,000/mm3
   * Total bilirubin < 2.5 X institutional upper limit of normal
   * AST, ALT < 2.5 X institutional upper limit of normal
   * Creatinine < 1.5 X institutional upper limit of normal
   * Normal cardiac function as determined by standard institutional methods
7. Women of child bearing potential must agree to use adequate contraception prior to study entry and for the duration of study.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Must have demonstrated resistance to steroids equivalent to >160mg/month of dexamethasone, 1g/month of prednisone, or 800mg/month of solumedrol, to insure the effects seen are from thymoglobulin and not the concomitant steroids.

Exclusion Criteria:

1. Receiving any other investigational agents.
2. Receiving concurrent steroids with a dose equivalent of dexamethasone of > 200 mg/month, 1.25g/month of prednisone, or 1g/month of solumedrol.
3. Pregnant or nursing.
4. Active systemic infection considered opportunistic, life threatening or clinically significant at the time of treatment.
5. Severe concurrent disease, including severe insulin-dependent diabetes, uncontrolled hypertension, transient ischemic attacks, uncontrolled symptomatic coronary artery disease, or symptomatic CNS involvement or psychiatric illness/social situations that would limit compliance with study requirements.
6. History of other malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast unless the subject has been off treatment and free from disease for > 3 years.
7. Weight of <100 kg to avoid exceeding maximum allowed steroid dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and dose limiting toxicity of thymoglobulin in multiple myeloma patients. | End of cycle 1 (DLT) and approximately 16 months after start of treatment (MTD)

SECONDARY OUTCOMES:
Determine the overall response rate (CR+PR) of patients with relapsed or refractory multiple myeloma treated with thymoglobulin | Day 14, Day 28 and Day 56
To determine the time to response, duration of response, and time to progression and overall survival | Until disease progression but no less than 30 days after end of treatment
To determine the safety and tolerability of thymoglobulin | 30 days after end of treatment
Assess the changes in lymphocyte apoptosis signaling in treated patients | Day 28 and Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington Universtiy in St. Louis
Locations (1):
- Washington Unvierstiy in St. Louis, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu